CLINICAL TRIAL: NCT02891694
Title: Metalloproteinases and Recurrent Corneal Erosion Syndrome
Acronym: MERCURE
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: EGN_2016_8
Record Dates: First submitted 2016-08-25; First posted 2016-09-07 (Estimated); Last update posted 2020-12-10 (Actual); Status verified 2020-12

CONDITIONS: Recurrent Corneal Erosion Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- recurrent corneal erosion
  Interventions: Other: in vitro immuno-histo-chemical analysis of corneal epithelium
- control patients (refractive surgery)
  Interventions: Other: in vitro immuno-histo-chemical analysis of corneal epithelium

INTERVENTIONS:
Other: in vitro immuno-histo-chemical analysis of corneal epithelium

SUMMARY:
Recurrent corneal erosion (RCE) syndrome can be observed either in the context of a dystrophy of the basement membrane or following corneal trauma. This syndrome is characterized by recurrent episodes of ocular pain more or less associated with localized separations between the outer epithelium and the epithelial basal lamina (basement membrane) because of anchorage abnormalities between these two corneal layers. This could be the result of an increased expression of metalloproteinases cleaving the hemidesmosomes which anchor epithelium to the basement membrane.

The investigators hypothesis is that episodes of RCEs are favored by a hyper- expression of matricial metalloprotease 9 (MMP-9) induced by EMMPRIN and Galectin-3. The identification of such induction could lead to development of therapeutics inhibiting EMMPRIN and Galectin- 3 in the RCE syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Recurrent Corneal Erosion Syndrome, with - failure of medical treatment and therapeutic photokeratectomy scheduled
* Photorefractive surgical keratectomy (control patients)

Exclusion Criteria:

* Opposition to participation in the study
* Known pregnancy or breast-feeding patient
* No medical insurance coverage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Recurrent Corneal Erosion Syndrome and control patients (undergoing photorefractive surgical keratectomy)
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2016-12-02 (Actual); Primary Completion 2020-06-26 (Actual); Study Completion 2020-11-26 (Actual)

PRIMARY OUTCOMES:
expression of the Extracellular Matrix Metalloproteinase Inducer (EMMPRIN) in epithelial cells | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Eric GABISON, MD, PhD, Principal Investigator — Fondation OPH A de Rothschild
Locations (1):
- Fondation Opthalmologique A de Rothschild, Paris, France